CLINICAL TRIAL: NCT07206784
Title: Understanding the Public Impact on Dengue Vaccination Strategies in Yunnan Province, China: A Dynamic Transmission Modeling Study
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yao, Ye, Associate Professor of Fudan University, Fudan University
Other Study IDs: IRB00002408 & FWA00002399
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Dengue Vaccination Strategy Evaluation; Transmission Modeling of Dengue; Public Health Impact of Vaccination

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a collaboration between the School of Public Health at Fudan University and the Xishuangbanna Center for Disease Control and Prevention in Yunnan Province, China. It aims to evaluate the public health impact of dengue vaccination strategies using dynamic transmission models. By simulating different vaccination scenarios, the study will assess the potential effectiveness and public health benefits of dengue vaccine introduction, providing scientific evidence to support local dengue prevention and control efforts.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Jinghong City, Xishuangbanna Prefecture
* Aged 3 years and above
* Able and willing to provide informed consent (or have legal guardian consent for minors)
* Available for blood sample collection between May and August 2025

Exclusion Criteria:

* Individuals with bleeding disorders or other contraindications to blood draw
* Individuals currently diagnosed with acute dengue infection

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Jinghong City, Xishuangbanna Prefecture, aged 3 years and older, selected across eight age groups for serological investigation of dengue virus exposure.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Dengue Virus Serological Response (IgM and IgG Antibody Levels) | From blood sample collection to the completion of laboratory analysis of dengue serology, serotype identification, and whole genome sequencing, from May to August 2025

CONTACTS AND LOCATIONS:
Locations (1):
- Xishuangbanna Center for Disease Control and Prevention, Jinghong, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided